CLINICAL TRIAL: NCT03969433
Title: Longitudinal Study for the Development of Innovative Wearable Tools for Foetal Wellbeing Monitoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bloom Technologies (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BEATLE
Record Dates: First submitted 2019-05-28; First posted 2019-05-31 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Foetal Wellbeing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase I (Experimental): Data collections are performed with TMSi Porti system and CTG (reference)
  Interventions: Device: TMSi Porti
- Phases II-III-IV (Experimental): Data collections are performed with the Bloomlife sensor and CTG (reference)
  Interventions: Device: Bloomlife sensor

INTERVENTIONS:
Device: TMSi Porti — Data collections
  Arms: Phase I
Device: Bloomlife sensor — Data collections
  Arms: Phases II-III-IV

SUMMARY:
The purpose of this study is to support the development of a new generation of the Bloomlife sensor, enabling continuous monitoring of foetal wellbeing.

Data is collected in four Phases, with different experimental setups. Recordings with investigational and reference devices are performed on the subjects, at different gestational ages.

The collected data is used for developing algorithms for the extraction of parameters descriptive of foetal wellbeing.

Clinical information related to subjects' pregnancy and foetal health is also collected.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant
* Gestational age of at least 20 weeks
* Singleton pregnancy
* Willingness to participate in the study

Exclusion Criteria:

* Multiple pregnancy
* Implanted pacemaker or any other implanted electrical device
* History of allergies to silicone-based adhesives

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2021-06-24 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Accuracy and reliability in the detection of foetal heart rate | Throughout the subject's participation in the study, from inclusion until delivery
  Foetal heart rate is extracted from the collected electrophysiological data and compared to the reference
Accuracy and reliability in the detection of foetal movements | Throughout the subject's participation in the study, from inclusion until delivery
  Foetal movements are detected from the collected sensor data and compared to the reference

CONTACTS AND LOCATIONS:
Overall Officials: Wilfried Gyselaers, MD, PhD, Principal Investigator — Ziekenhuis Oost-Limburg
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: Undecided